CLINICAL TRIAL: NCT04740996
Title: A Prospective Registration Study of Pembrolizumab in the First Line Therapy for PD-L1 CPS≥20 Recurrent or Metastatic Head and Neck Squamous Cell Carcinoma in China
Brief Title: Study of Pembrolizumab in the First Line Therapy for R/M HNSCC in China
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shi Yuankai (Unknown)
Responsible Party: Sponsor-Investigator, Shi Yuankai, Director, Head of Oncology, Chief physician, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Other Study IDs: NCT123
Record Dates: First submitted 2021-02-02; First posted 2021-02-05 (Actual); Last update posted 2022-02-07 (Actual); Status verified 2022-02

CONDITIONS: Head and Neck Squamous Cell Carcinoma
Keywords: Head and Neck Cancer; immune therapy; Pembrolizumab
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Head and Neck Neoplasms | interventions — pembrolizumab

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Pembrolizumab — Pembrolizumab (formerly lambrolizumab, brand name Keytruda) is a humanized antibody used in cancer immunotherapy. This includes to treat melanoma, lung cancer, head and neck cancer, Hodgkin lymphoma, and stomach cancer.
  Other Names: keytruda

SUMMARY:
This trial is main evaluate the efficacy and safety of pembrolizumab in the first-line treatment of Chinese patients with recurrent or metastatic head and neck squamous cell carcinoma with PD-L1 CPS≥20.

DETAILED DESCRIPTION:
This trial is a single-center, prospective phase II clinical study, which mainly evaluates the efficacy and safety of first-line treatment with pembrolizumab in patients with recurrent and/or metastatic head and neck squamous cell carcinoma with PDL1 CPS≥20 in China.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily sign a written informed consent before screening;
2. Male or female, aged ≥18 years old;
3. ECOG physical status score 0-1 points;
4. Head and neck squamous cell carcinoma (HNSCC) confirmed by histology or cytology, the primary site is oral cavity, oropharynx, hypopharynx or larynx;
5. Recurrent and/or metastatic HNSCC without indications for local radical treatment;
6. According to the evaluation criteria for the efficacy of solid tumors (RECIST version 1.1), there is at least one measurable lesion. For lesions that have received radiotherapy in the past, they can only be selected as the disease if there is a clear disease progression 3 months after the end of radiotherapy. Target lesion
7. PD-L1 immunohistochemical detection of tumor tissue samples with CPS≥20;
8. The expected survival period exceeds 3 months;
9. The main organs function normally, that is, they meet the following standards:

   i. Routine blood test (not receiving blood transfusion, erythropoietin (EPO), granulocyte colony stimulating factor (G-CSF) or granulocyte-macrophage colony stimulating factor (GM-CSF) within 14 days before the screening examination) : Neutrophils ≥1.5×109/L, platelets ≥100×109/L, hemoglobin ≥90g/L; ii. Liver function: alanine aminotransferase (ALT) and aspartate aminotransferase (AST), ALT and AST≤3×ULN for those without liver metastasis, ALT and AST≤5×ULN for those with liver metastasis; total bilirubin (TBIL)≤ 1.5×ULN (Patients with Gilbert syndrome, ≤3×ULN); iii. Renal function: serum creatinine (Cr) ≤1.5×ULN or creatinine clearance (Ccr) ≥50ml/min; iv. Coagulation function: activated partial thromboplastin time (APTT), international normalized ratio (INR), prothrombin time (PT)≤1.5×ULN;
10. Heart echocardiogram: left ventricular ejection fraction (LVEF) ≥50%;
11. Women should agree to use contraceptive measures (such as intrauterine device [IUD], contraceptives or condoms) during the study period and 6 months after the end of the study; the blood pregnancy test is negative within 7 days before the study is enrolled, And must be a non-lactating patient; men should agree to patients who must use contraception during the study period and within 6 months after the end of the study period.

Exclusion Criteria:

1. Patients who are suitable for local treatment and are willing to local treatment;
2. Have received systemic chemotherapy, but does not include chemotherapy for locally advanced disease as a part of multimodal treatment (the end of this treatment must be more than 6 months from the first trial drug); Note: Multimodal treatment includes induction chemotherapy, concurrent radiotherapy and chemotherapy and adjuvant chemotherapy.
3. Locally advanced head and neck squamous cell carcinoma multimodal treatment is completed within 6 months of disease progression;
4. Have previously been immunized with anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137 or anti-CTLA-4 antibodies or any other antibodies or drugs that target T cell co-stimulation or immune checkpoint pathways treatment;
5. Other malignant tumors occurred within 5 years or at the same time during the current period, except for cured cervical carcinoma in situ, non-melanoma skin cancer, or other tumors/cancers that have undergone radical treatment and have no signs of disease for at least 5 years;
6. Received cetuximab treatment within 6 months before the first administration;
7. According to the standard of common adverse event term (NCI CTCAEv5.0), peripheral neuropathy has been ≥2 grade;
8. Accompanied by known active central nervous system metastasis (CNS) and/or cancerous meningitis: Subjects with brain metastases who have received previous treatment can participate in the study, provided that they are clinically stable for at least 2 weeks and there are no new or expanded ones Evidence of brain metastases, and steroids were stopped 14 days before study drug administration. Stable brain metastases in this definition should be determined before the first administration of the study drug. Subjects with asymptomatic brain metastases (that is, no neurological symptoms, no corticosteroids, and no lesions> 1.5 cm) can participate, but they need to have regular brain imaging examinations as the disease site;
9. Subjects who have not recovered from any acute effects of previous surgery, chemotherapy or radiotherapy, that is, subjects who have not fallen to ≤1 (NCI CTCAEv5.0) (except for hair loss). If the nutritional status is stable, allow the chronic late toxicity (pharyngeal/laryngo toxicity, dry mouth, abnormal speech, swallowing, etc.) from previous radiotherapy and/or surgery;
10. Any component of the studied drug or preparation has caused severe allergic reactions, including known severe allergic reactions to other monoclonal antibodies (NCI CTCAEv5.0≥3);
11. Have received anti-tumor drug therapy (such as chemotherapy, hormone therapy, immunotherapy, antibody therapy, radiotherapy, etc.) 4 weeks or 4 weeks before the first administration, except for palliative radiotherapy for bones to relieve pain;
12. Chinese herbal medicines or proprietary Chinese medicines that have received anti-tumor treatment ≤1 week before the first administration;
13. Have received major surgery within 4 weeks before the first administration or are expected to undergo major surgery during the study period;
14. Immunosuppressive drugs need to be used 2 weeks before the first administration or within 2 weeks or during the study period, except for the following conditions:

    1. Intranasal, inhaled, topical steroid or topical steroid injection (such as intra-articular injection);
    2. Physiological dose of systemic corticosteroids (≤10mg/day prednisone or equivalent dose);
    3. Short-term (≤7 days) use of steroids to prevent or treat non-autoimmune allergies Sexual disease
15. Subjects who are known to have active or have a history of autoimmune diseases that are likely to relapse (such as systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, autoimmune thyroid disease, Patients with multiple sclerosis, vasculitis, glomerulitis, etc.), or high-risk (such as receiving an organ transplant and requiring immunotherapy). However, the following patients are allowed to join the group: patients with type I diabetes who are in stable condition after using a fixed dose of insulin; autoimmune hypothyroidism who only needs hormone replacement therapy; skin diseases that do not require systemic treatment (such as eczema, which occupies body surface Less than 10% of skin rashes, psoriasis without ophthalmological symptoms, etc.);
16. Subjects with known history of interstitial lung disease, history of non-infectious pneumonia, or high suspicion of interstitial lung disease; subjects who have previously had drug-induced or radiation non-infectious pneumonia but asymptomatic are allowed to enter group;
17. History of infection with human immunodeficiency virus (positive HIV test), or other acquired or congenital immunodeficiency diseases, or history of organ transplantation, or history of stem cell transplantation;
18. At the time of screening, the hepatitis B or C virology test meets any of the following:

    1. HBsAg is positive and the titer of hepatitis B virus deoxyribonucleic acid (HBV DNA) in peripheral blood is ≥104 copies/ml or ≥2000 IU/ml;
    2. HCV antibody is positive, and HCV-RNA is higher than the detection limit of the analysis method;
19. Within 2 weeks or 2 weeks before the first administration, the subject has an active infection or uncontrollable infection that requires systemic treatment (except simple urinary tract infection or upper respiratory tract infection);
20. Live virus vaccine has been vaccinated within 4 weeks before the first dose. Allow seasonal influenza vaccination without live virus;
21. Serous effusion (such as pleural effusion and ascites) with clinical symptoms that require clinical intervention or stable time less than 4 weeks;
22. Known to be accompanied by serious medical diseases, such as cardiac dysfunction of grade III and above (New York Heart Association [NYHA]), cardiovascular diseases such as ischemic heart disease (such as myocardial infarction or angina), or the first administration A history of myocardial infarction within the first 3 months, poorly controlled diabetes (fasting blood glucose ≥10mmol/L) or poorly controlled hypertension (systolic blood pressure ≥160mmHg and/or diastolic blood pressure ≥100mmHg) after drug treatment;
23. Medical or psychiatric history or laboratory abnormality history that may interfere with the interpretation of results;
24. The subject is currently enrolled in another research device or research drug study, or the time away from stopping other research drugs or research devices is less than or equal to 4 weeks;
25. The subject is known to be addicted to alcohol or drugs;
26. The researcher believes that the subject has other conditions that may affect its compliance with the protocol and the evaluation of the research indicators, and it is not suitable for the subjects to participate in the research.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with recurrent and/or metastatic head and neck squamous cell carcinoma who are about to receive advanced first-line treatment.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2021-02-04 (Actual); Primary Completion 2024-02 (Estimated); Study Completion 2024-02 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | 1 year
  To evaluate the objective response rate (ORR, RECIST standard 1.1 evaluation) of pembrolizumab in the first-line treatment of Chinese patients with recurrent and or metastatic head and neck squamous cell carcinoma with PDL1 CPS≥20
survival time (OS) | 1year
  To evaluate the survival time (OS) of pembrolizumab in the first-line treatment of Chinese patients with recurrent and or metastatic head and neck squamous cell carcinoma with PDL1 CPS≥20

SECONDARY OUTCOMES:
objective response rate(ORR) | 1 year
  To evaluate the objective response rate of pembrolizumab in the first-line treatment of Chinese patients with recurrent and or metastatic head and neck squamous cell carcinoma with PDL1 CPS≥20 (ORR, iRECIST standard evaluation)
disease control rate (DCR) | 1 year
  To evaluate the disease control rate (DCR) of pembrolizumab in the first-line treatment of Chinese patients with recurrent and or metastatic head and neck squamous cell carcinoma with PDL1 CPS≥20
duration of response (DOR) | 1 year
  To evaluate the duration of response (DOR) of pembrolizumab in the first-line treatment of Chinese patients with recurrent and or metastatic head and neck squamous cell carcinoma with PDL1 CPS ≥ 20
progression-free survival (PFS, PFS2) | 1 year
  To evaluate the progression-free survival (PFS, PFS2) of patients with recurrent and or metastatic head and neck squamous cell carcinoma with PDL1 CPS ≥ 20 in the first-line treatment of Pembrolizumab;

OTHER OUTCOMES:
TMB, T cell gene expression | 3 year
  Correlation between the results of TMB and inflammatory T cell gene expression profiles in tumor tissues of baseline patients and the efficacy and prognosis.

CONTACTS AND LOCATIONS:
Overall Officials: Yuankai Shi, MD, Principal Investigator — Cancer Institute/Hospital, Chinese Academy of Medical Sciences & Peking Union Medical College
Locations (1):
- Cancer Institute/Hospital, Chinese Academy of Medical Sciences & Peking Union Medical College, Beijing, China

IPD SHARING:
Plan to Share IPD: No